CLINICAL TRIAL: NCT02271685
Title: Estimation and Accuracy in Sound Task Perceived to be Medically Diagnostic
Brief Title: Sound Estimation and Accuracy Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, PhD Candidate, Carnegie Mellon University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: HS14-553
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's; Alzheimer Disease
Keywords: Diagnostic Information; Risk Perception
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Overestimate Parkinson's (Experimental): People are told that overestimates on the sound estimation task are associated with being healthy and having a low risk of Parkinson's disease, whereas those who are accurate are more likely to develop the disease later in life.
  Interventions: Other: Instructions about Overestimates; Other: Instructions about Parkinson's
- Overestimate Alzheimers (Experimental): People are told that overestimates on the sound estimation task are associated with being healthy and having a low risk of Alzheimers disease, whereas those who are accurate are more likely to develop the disease later in life.
  Interventions: Other: Instructions about Overestimates; Other: Instructions about Alzheimers
- Underestimate Parkinson's (Experimental): People are told that underestimates on the sound estimation task are associated with being healthy and having a low risk of Parkinson's disease, whereas those who are accurate are more likely to develop the disease later in life.
  Interventions: Other: Instructions about Parkinson's; Other: Instructions about Underestimates
- Underestimate Alzheimers (Experimental): People are told that underestimates on the sound estimation task are associated with being healthy and having a low risk of Alzheimers disease, whereas those who are accurate are more likely to develop the disease later in life.
  Interventions: Other: Instructions about Underestimates; Other: Instructions about Alzheimers

INTERVENTIONS:
Other: Instructions about Overestimates — Participants are told that overestimating the duration of sounds are associated with low disease risk.
  Arms: Overestimate Alzheimers; Overestimate Parkinson's
Other: Instructions about Parkinson's — Participants are told that the task is about risk of Parkinson's disease.
  Arms: Overestimate Parkinson's; Underestimate Parkinson's
Other: Instructions about Underestimates — Participants are told that underestimating the duration of sounds are associated with low disease risk.
  Arms: Underestimate Alzheimers; Underestimate Parkinson's
Other: Instructions about Alzheimers — Participants are told that the task is about risk of Alzheimers disease.
  Arms: Overestimate Alzheimers; Underestimate Alzheimers

SUMMARY:
Participants will be assigned to complete computerized estimation tasks for which there is a component of accuracy, such as estimating the duration of sounds. Participants will be told that the task is used as an early diagnostic tool to detect those at risk for a medical condition (e.g., Parkinson's disease, Alzheimer's disease). Instructions will be given to participants telling them that accuracy on the task is associated with the disease, whereas those who are not at risk of the disease tend to either overestimate or underestimate the duration of the sounds. The investigators examine whether such instructions about the purpose and diagnosticity of the tasks biases participants' responses to the tasks, leading them to purposefully be more inaccurate in their estimates.

DETAILED DESCRIPTION:
Participants will be assigned to complete computerized tasks for which there is a component of accuracy, such as estimating the length, in time, of sounds. Participants will be told that the task is used as an early diagnostic tool to detect those at risk for a medical condition (e.g., Parkinson's disease, Alzheimer's disease). Instructions will be given to participants telling them that accuracy on the task is associated with the disease in question, whereas those who are not at risk of the disease tend to either overestimate or underestimate the duration of the sounds. The investigators examine whether such instructions about the purpose and diagnosticity of the tasks biases participants' responses to the tasks. The investigators collect additional survey measures as statistical controls and potential explanatory variables for variation in the performance on the tasks, and also test whether financial incentives for accuracy on these tasks improve the accuracy of responses to these tasks.

Following the task, all participants will be told that the tasks used are actually NOT diagnostic of the diseases in question, and that deception was used to learn how people respond to instructions about how a task can be used for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Able to access tasks on computer
* Able to hear sounds played on computer

Exclusion Criteria:

* Computer speakers absent or not functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time Estimate | 30 minutes
  The estimate of the length of time elapsed during the sound file

SECONDARY OUTCOMES:
Time Generation | 30 minutes
  The length of time selected for the sound file to run by participants in a secondary task
Perceived Risk of Disease | 30 minutes
  Scale question asking participants their perceived risk of having the diseases in the study

CONTACTS AND LOCATIONS:
Overall Officials: Eric M VanEpps, MS, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States